CLINICAL TRIAL: NCT04289714
Title: A Feasibility Study to Assess Novel Electronic Monitoring Devices (NEMD) for Monitoring Adherence in Children With Asthma
Brief Title: Novel Electronic Monitoring Devices (NEMD) to Monitor Adherence in Children With Asthma
Acronym: NEMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Asthma UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 239759
Record Dates: First submitted 2020-02-21; First posted 2020-02-28 (Actual); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Asthma in Children
Keywords: Asthma; Children; Adherence; Electronic Monitoring devices (EMD); Inhalers; Inhaled medication
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Feasibility Pragmatic randomisation
Masking Description: Pragmatic randomization based on inhaled medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- R-DOT (Experimental): Remote Directly Observed Therapy
  Interventions: Device: Novel Electronic Monitoring Device
- Haillie (Experimental): Smartinhaler Haillie
  Interventions: Device: Novel Electronic Monitoring Device
- Rafi-tone/INCA (Experimental): Rafi-tone with Flo-tone /INCA
  Interventions: Device: Novel Electronic Monitoring Device

INTERVENTIONS:
Device: Novel Electronic Monitoring Device — Four Novel electronic Monitoring Devices were trialled

SUMMARY:
This is a feasibility study to assess novel electronic monitoring devices for monitoring adherence in children with asthma who are on inhaled corticosteroids (ICS)

It is a mixed method (quantitative and qualitative) open label, pragmatic randomised feasibility study with two main aims:

1. To assess the feasibility of 4 novel electronic monitoring devices in children aged 6-16 years with asthma, in terms of usability and acceptability by patients/ guardians and healthcare professionals (qualitative study)
2. To evaluate the accuracy of these devices and assess whether they impact on asthma control (quantitative study).

The duration of study is 16 weeks.

DETAILED DESCRIPTION:
This was an open label, block randomised (10 in each block), mixed method (quantitative and qualitative) study to be conducted for a period of up to 16 weeks

Children aged between 6-16 years with asthma attending the paediatric respiratory difficult asthma clinic will be recruited into the study and randomly allocated to one of three arms using block randomisation matched for age and size of group. Children will be assigned to trial one of the following four NEMD's to be tested:

1. Block 1 (10): Smart-inhaler Plus™ (Adherium, New Zealand)

   • This measures inhalation usually flow sensors and is the next generation of a currently commercially available EMD
2. Block 2a (5) : Flo-Tone (Clement Clarke, UK) plus Rafi-tone, acoustic enabled Smartphone App (clin-e-cal, UK) for children aged 6 - 11 years • The Flo-Tone attaches to a Metered Dose Inhaler (MDI) and makes a sound when the inhaler is used correctly. Rafi-tone is a Smartphone App that detects the sound and activates a game The game is aimed at younger children and therefore children aged 6 - 11 years will be randomised to this block.

Block 2b (5) : Inhaler Compliance Assessment (INCA™) device (INCA, Ireland)

* This is an audio recording device which attaches to a Discus dry powder inhaler. Analysis of the digital audio recordings enables objective assessment of inhaler use and technique. As it can only be used with a Discus only children ≥ 12 years will be randomised to this block

  3. Block 3: Video and Remote Directly Observed treatment (rDOT)
* Children are filmed on a Smartphone using their inhaler. The clip is then automatically uploaded via a Smartphone App (Continga, UK) and reviewed by a Clinical Nurse Specialist to ensure inhaler technique is correct.

Recruitment :

The aim was to recruit 30 children into the study; 10 per block, and 5 per block aged 6-11 years and 5 aged 12-16 years for the INCA/Rafi-tone arm. However, due to low number of participants completing the study, ethics approval was sought to extend the study. As a result 35 participants were recruited at the end of the study period.

Visit 1:Novel electronic monitoring device (NEMD) issued Routine clinical care assessments will be carried out at the end of the study period as below, including asthma control test (ACT) or the childhood asthma control test (cACT), exhaled nitric oxide (FeNO) and spirometry (FEV1 and BDR) .

Patient/parent/Carer will be invited to take part in the study. Information regarding the study and its objectives will be communicated to the Patient/parent/carer in both oral and written form using patient information leaflets.

All children will be issued with a novel electronic monitoring device which will be attached to the child's usual inhaler or require an app on their mobile phone as described above. Parents and children will be provided information and advice on the use of the novel electronic monitoring device and asked to conduct up to 16 weeks of home monitoring using their allocated NEMD on their first visit.

Information on how to contact the team in case of any problems will be related to the participant in both oral and written form.

The data will be stored electronically and downloaded at the next clinic visit. Contact by telephone will be made at day 7-14 to ensure that the device is working and to answer any other queries then at week 6-7 to determine if the device is being used appropriately and to answer any related questions.

Week 1 - for the rDOT arm, adherence data will be downloaded to check for consistencies in inhaler technique. If inhaler technique is inaccurate, the participants will be called by the respiratory nurse specialists to advise on correct technique. This will be documented as part of the data collection.

Week 4 - All devices, adherence data will be downloaded and checked to ensure that the devices are working correctly.

Visit 2: up to 12 weeks of adherence data collection Routine clinical care assessments will be carried out at the end of the study period as below, including asthma control test (ACT) or the childhood asthma control test (cACT), exhaled nitric oxide and spirometry (FEV1 and BDR) .

Adherence data will downloaded at the end of the study period and stored electronically.

Visit 3: Focus group or one to one interviews The participants and their carers will be invited to a face to face focus group interview, or a one to one interview, depending on their availability at the end of the study period. The focus group and one to one interviews will utilise a semi structured questionnaire, to provide qualitative feedback on the acceptability and usability of the devices.

A separate focus group meeting will also be conducted with the paediatric respiratory nurses who are part of the Multi disciplinary Team (MDT) to assess their views on the devices used as they routinely provided all asthma devices and are also involved in downloading data from other devices that the investigators would use as part of routine care (smart-inhaler). They will also be consented to take part in the study Where possible a second researcher from University College London (UCL), Christina Pearce will sit in the focus groups discussion and interviews to ensure there is no bias.

The conversations from the focus group and one to one interviews will be transcribed and coded into themes. The investigators will utilise an external company for transcribing the conversations called 1st Class.

Analysis

Qualitative:

The focus group and one to one interviews will be audio recorded, transcribed and put into themes to conduct an inductive thematic analysis. 25% of the transcripts (8) will be double coded by an independent researcher from UCL, Dr Amy Chan, experienced in qualitative research to ensure that the correct themes have been used and to ensure that there is no bias.

The focus group and one to one interviews will be used to assess the usability and acceptability of the devices

Quantitative:

The amount of usable data from each device will be quantified and compared. This will provide data on the perceived accuracy of the device.

The quantitative and qualitative results will be amalgamated and an evidence report prepared to assess the feasibility of each device.

An expert panel will be convened to select the most appropriate device to take forward to a larger randomised controlled trial to assess the impact of the device on adherence in children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from parents/guardian/adolescents and/or assent from the child.
* Children aged between 6-16 years with a diagnosis of asthma attending the Royal Brompton and Harefield Difficult asthma clinic.
* Children on inhaled cortico-steroids
* Parents/ young person has a mobile phone which can download apps
* Paediatric respiratory nurses working in the difficult asthma team at Royal Brompton Hospital.

Exclusion Criteria:

* Unable to provide consent
* As a result of medical interview, physical examination or screening investigation the physician responsible considers the child unfit for the study.
* Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures
* Children under the age of 6 years.
* Children not on inhaled cortico-steroid
* It is not anticipated that any children will be pregnant, however, if they are they will not be included in the study

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise Fleming, MD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be shared in a publication format.
Supporting Information: ICF
Time Frame: 6 months from publication
Access Criteria: For publication purposes by the Principal investigator and the study team

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The initial recruitment total was 30, however, due to low number of participants completing the study, ethics approval was sought to extend the study. As a result 35 participants were recruited at the end of the study period.
Period: Overall Study
Arm/Group | R-DOT | Haillie | Rafi-tone/INCA
Started | 14 | 11 | 10
Completed | 8 | 6 | 4
Not Completed | 6 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R-DOT | Haillie | Rafi-tone/INCA | Total
Number analyzed (Participants) | 14 | 11 | 10 | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [7 to 16] | 13.5 [11 to 15] | 12 [9 to 14] | 13 [7 to 16]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number analysed are differ from the number at baseline as these are the ones that completed the study
  Participants
    number analyzed (Participants) | 8 | 6 | 4 | 18
    Female | 4 | 5 | 2 | 11
    Male | 4 | 1 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Acceptability Using Semi Structured Questionnaires in Focus Groups and Interviews
Description: Number of participant interviewed in focus groups and interviews
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | R-DOT | Haillie | Rafi-tone/INCA
Number analyzed (Participants) | 8 | 6 | 4
Participants | 7 | 4 | 3

2. Primary Outcome: Number of Themes Generated by Participants Regarding Usage of the Devices
Description: The Primary outcome measure is largely qualitative and based on collective themes. As a result there are no numerical measurements that differ each of the devices. In terms of accuracy of each device adherence data was collected but differs for each device depending on its functionality
Time Frame: 16 weeks
Population: Number of discussion themes generated by participants regarding the usage of the devices
Measure: Number; unit: ber of discussion themes generated by pa
Units Other Than Participants: Number of themes generated
Arm/Group | R-DOT | Haillie | Rafi-tone/INCA
Number analyzed (Participants) | 7 | 4 | 3
Number analyzed (Number of themes generated) | 4 | 4 | 4
ber of discussion themes generated by pa | 4 | 4 | 4

3. Secondary Outcome: Adherence to Inhaled Medication
Description: Percentage adherence to inhaled corticosteroids
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Percentage adherence to inhaled corticos
Arm/Group | R-DOT | Haillie | Rafi-tone/INCA
Number analyzed (Participants) | 8 | 6 | 4
Percentage adherence to inhaled corticos | 72 (13) | 65 (19) | 87 (7)

ADVERSE EVENTS:
Time Frame: AE data was not collected due to it being an observational study and no AE's were anticipated.
Description: No AE's were expected and AE's were not monitored for this reason.
Arm/Group | R-DOT | Haillie | Rafi-tone/INCA
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The numbers completing in each arm was small to calculate robust quantitative analysis, however, it was a sufficient size for qualitative analysis which was the primary aim of the study. The study period was extended due to low completion rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT04289714/Prot_SAP_000.pdf